CLINICAL TRIAL: NCT05333939
Title: Investigating the Effect of Moringa Oleifera Leaf Powder on Breastmilk Quantity and Quality: a Double Blinded Randomized Placebo-controlled Trial
Brief Title: Moringa Supplementation for Improved Milk Output
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kentucky (Other)
Collaborators: University of Idaho (Other)
Responsible Party: Principal Investigator, Suzanna L Attia, Assistant Professor, University of Kentucky
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PED-22-MORINGA
Record Dates: First submitted 2022-03-28; First posted 2022-04-19 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Breastfeeding
Keywords: maternal and child health
MeSH Terms: conditions — Breast Feeding | interventions — flocculant protein MO 2.1, Moringa oleifera; Starch

STUDY DESIGN:
Intervention Model Description: placebo controlled randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Moringa (Experimental): 4 g moringa leaf powder in green capsules divided into 4 capsules twice daily x 7 days
  Interventions: Dietary Supplement: Moringa leaf powder
- Control (Placebo Comparator): comparable weight green capsules with cornstarch divided into 4 capsules twice daily x 7 days
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Moringa leaf powder — capsule ingestion
  Other Names: moringa oleifera
  Arms: Moringa
Other: Placebo — capsule ingestion
  Other Names: cornstarch
  Arms: Control

SUMMARY:
The overall objective is to obtain preliminary data on the effect of Moringa oleifera leaf supplementation (moringa) at 4g daily for four weeks compared to placebo to improve human milk quantity and quality and infant health. Hypothesis: Four grams of moringa daily by mouth compared to placebo will increase breastmilk output and percent of mother's own milk consumed by infant.

ELIGIBILITY:
Mom

YES:

* willing to breastfeed or pump for one week
* willing to complete study activities (at minimum measure 24 hour pumped volume at start and end of capsules, take capsules daily, and answer questions)
* has access to breastpump (in hospital and/or home)
* English speaking
* 18 years or older
* Gave birth between 2-6 weeks prior to study start

NO:

* taking metoclopramide (trade name Reglan) currently or within 2 weeks of enrollment
* taking moringa regularly or within 2 weeks of enrollment
* breast surgery (amplification, reduction, or other)
* breast condition: Insufficient Glandular tissue
* unprescribed or street drug use at any point in pregnancy, or enrolled in rehab program or receiving addiction therapy
* refuses to take 4 capsules twice daily within 2 days of study start
* wishes to withdraw within 2 days of study start

Infant

YES:

* 28-36 and 7 weeks gestation (ie 37 weeks is too old)
* 2-6 weeks old
* singleton birth

NO:

· any condition where breastmilk is clinically contraindicated

Min Age: 0 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2024-08-03 (Actual); Study Completion 2024-08-03 (Actual)

PRIMARY OUTCOMES:
Milk output | 7 days
  24 hour milk output at 7 days

SECONDARY OUTCOMES:
% mother's own milk consumed by infant | 7 days
  % of mother's own milk (over total enteral nutrition) consumed by infant at 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Suzanna Attia, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No